CLINICAL TRIAL: NCT06910605
Title: Exploring Parameters of Driving Simulation in Relation to Drug Holidays in ADHD Patients
Acronym: DS-ADHD1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefan Lakämper (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other); Swiss Federal Institute of Technology in Zurich (ETHZ) (Unknown)
Responsible Party: Sponsor-Investigator, Stefan Lakämper, Dr. rer. nat. , Head Research & Research Development, Division of TRaffic Medicine, Institute for Forensic Medicine, University of Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DS-ADHD1
Record Dates: First submitted 2025-03-14; First posted 2025-04-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; Driving Simulator Performance; ADHD; Driving Behavior; Driving Ability
Keywords: driving simulation; driving performance; eye tracking; EEG-recording; stimulant treatment; drug holidays
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Treatment Interruption; Fumigant 93

STUDY DESIGN:
Intervention Model Description: monocentric, within-subjects, observer-blinded cross-over trial (within-subject randomized crossover trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: M-M-D (Experimental): stimulant-treated ADHD-affected participants will perform test sequence first in medicated state (M), then again in medicated state (M), then during "drug holidays" (D).
  Interventions: Drug: "drug holidays" (D)
- Group 2: M-D-M (Experimental): stimulant-treated ADHD-affected participants will perform test sequence first in medicated state (M), then during "drug holidays" (D), then again in medicated state (M).
  Interventions: Drug: "drug holidays" (D)

INTERVENTIONS:
Drug: "drug holidays" (D) — Participants omit three consecutive daily doses of ADHD-medication (stimulant).

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) or syndrome (ADHS) is a symptomatically defined condition that - if untreated - is linked to a significantly increased risk of traffic accidents. In a recent umbrella review, where data from reviews and meta-analyses on 21.142.129 adults was assessed, a pooled prevalence of 3.1% of ADHD in adults was estimated. Considering that globally around 1.35 million people lose their lives and more than 50 million are suffering from injuries or disabilities due to road accidents, the fraction of car accidents caused by ADHD as a risk factor is considerable and needs to be addressed. This risk is largely presumed to be caused by an elevated level of inattentiveness in affected persons.

Compounds of different groups, which can be classified in stimulants - formulations of methylphenidate and amphetamine - and non-stimulants - atomoxetin, guanfacine and clonidine -, have been shown to be effective in alleviating negative effects of ADHD, including inattentiveness. Under well-established but individually managed medication regimes, affected individuals can consequently lead a largely "unirritated" life and are not subject to fundamental restriction with respect to driving anymore.

In children and adolescents, documented negative effects of stimulant medication include loss of appetite and decreased growth rates. It could however be shown that short-term interruptions (weekend, school holidays, and alike), introduced to alleviate aforementioned effects, do not affect the drug's beneficial effects in functional use (e.g., school). Such monitored medication breaks are often called "drug holidays" (D). They have become standard procedure in well-monitored treatment, predominantly including behavioral therapy.

Based on own experience in childhood and or hearsay, also a fraction of affected adults under stimulant medication expresses the desire to take drug holidays and "be themselves" from time to time. With the predominant fraction of medication being fast acting drugs in extended-release formulation and typical patients being not only highly compliant but also extremely informed and adherent, these so-called "drug holidays" are reported an accepted in therapeutically accompanied settings of adults by now.

However, while the overall positive effect of stimulant treatment on driving performance has been confirmed in a row of excellent on road- and/or simulation studies using integrated driving scores (IDS), so far there is no study available addressing the effect of drug holidays in adult drivers on driving performance. This represents a significant gap of evidence for both medical experts and affected.

The proposed study will address this gap by exploring parameters of driving simulation in relation to drug holidays in ADHD patients.

ELIGIBILITY:
Inclusion criteria:

* adult drivers
* ADHD-diagnosed, established ADHD-treatment only with stimulants
* known history of drug holidays based on own decision,
* at impaired eyesight with more than +/- 5 diopter or astigmatism
* contact lenses are required (for eye tracking)

Exclusion criteria:

* sensibility to motion sickness (kinetosis, dizziness etc. in 5 min screening drive)
* non-stimulant-treatment
* inability to understand the study procedure for linguistic or cognitive reasons
* professional drivers (if working during the study period)
* for women: pregnancy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Significant differences in IDS between conditions D and M | 0, x, x+3 days, with x≥ 4 days
  Primary outcome parameter IDS (Integrated Driving Score) will be calculated by summation of z-scores of typical driving parameters such as, for example, the standard deviation of lane position (SDLP), standard deviation of velocity (SDS) or number of inappropriate lane departures, ILD. IDS will be measured on day 0 (= baseline, Visit 1), on day x (with x≥4, Visit 2) and on day x+3 (Visit 3).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lakämper, Dr. rer. nat., Principal Investigator — University of Zurich; Kristina Keller, Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Division of Traffic Medicine, Institute of Forensic Medicine, University of Zurich,, Zurich, ZRH, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in peer-reviewed journals. Anonymized raw data will be made available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting after publication of study protcol and/or results
Access Criteria: upon request by mail